CLINICAL TRIAL: NCT07130812
Title: Breaking the Cycle of Low Back Pain: Blood Flow Restriction Training (BFR) as a Targeted Intervention for Rowers
Brief Title: Blood Flow Restriction Training as a Targeted Intervention for Rowers With Back Pain.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Everett Lohman, Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5250411
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Low Back Pain
Keywords: blood flow restriction
MeSH Terms: conditions — Low Back Pain | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Restriction Group (Active Comparator): Using blood flow restriction, participants partake in aerobic (rowing) and anaerobic (squats/deadlifts) exercises.
  Interventions: Other: blood flow restriction
- Non Blood Flow Restriction Group (Active Comparator): Participants partake in aerobic and anaerobic exercises without blood flow restrictions. The participants will use heavier loads in the anaerobic exercises.
  Interventions: Other: Heavy load resistance training

INTERVENTIONS:
Other: blood flow restriction — The SAGA blood flow restriction tourniquet system will be used for each training sessions for the rowers within the light load restriction group. The 4 inch-wide tourniquet will be applied to both upper thighs during the strength and endurance exercises. Tourniquet setting will be determined as the pressure needed to achieve 40-80% arterial occlusion to the extremity (as measured by the SAGA BFR unit). The SAGA units provides a consistent amount of pressure to the extremity throughout the ROM of the exercise. The settings will be determined at baseline and then recalibrated weekly.
  Arms: Blood Flow Restriction Group
Other: Heavy load resistance training — For the resistance prescription, rowers will do strengthening exercises at 70-80% 1 RM. Exercises will be performed in series following 6 sets by 5 reps, with 120 seconds of rest between sets for each exercise.
  Arms: Non Blood Flow Restriction Group

SUMMARY:
The purpose of this graduate student research study is to compare the effects of low-load blood flow restriction training (LL-BFR) and heavy-load training (HLT) in high-volume rowers with mild low back pain or recurrent low back pain (LBP), aiming to determine whether LL-BFR offers a safer yet equally effective alternative to HLT for enhancing performance and reducing risk of re-injury.

DETAILED DESCRIPTION:
Rowers will complete a web-based survey administered via administered via Google Forms for up to 15 minutes. Questions will address demographics, attendance adherence to rowing practice/races, a blood flow restriction pre-screening questionnaire, and the Orebro Musculoskeletal Pain Questionnaire (OMPQ) for LBP. Rowers will participate in a 2000-meter indoor rowing ergometer time trial to assess, technical fatigue, muscular fatigue, and performance. Muscular fatigue will be assessed through the use of Electromyography (EMG) collected via Noraxon Ultium electrodes and sensors on the hamstrings and quadriceps. Performance on the 2000-meter time trial will be determined by improvement of time to completion. Performance will be further assessed through a 1-repetition maximum (1RM) test for squat and deadlifts. Strength and endurance ratios will also be collected assessing hamstrings: quadriceps using an Asani tension dynamometer and abdominal endurance. Rowers will then be split into two groups (exercise and sham) through blocked randomization: light-load blood flow restriction training (LL-BFR) and heavy load training (HLT). Each LL-BFR session will include the following strength exercises at 20-30% of each participant's 1 RM: (1) Squats (Goblet/Back squat), (2) Deadlifts (Conventional/Romanian), (3) Side planks, (4) Plank, and (5) Bird-Dogs. The exercises will follow a 4-set structure: Set 1 with 30 repetitions, followed by three sets of 15 repetitions, with 30-second rests between each set. Participants will report their rating of perceived exertion (RPE) on a 1-10 scale, aiming to maintain an RPE of 7-8; load and occlusion pressure can be adjusted accordingly. The HLT will participate in the same exercises but under a different dosage of 6 sets and 5 reps at 60-80% 1 RM.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13-20 years old
* Currently active rower (training ≥3 days/week or 12 hours/week)
* Mild LBP with a low reactivity (<3/10) or recurring LBP within the past 18 months that has affected attendance to team practices/races.
* Able to complete a 2,000-meter rowing erg test

Exclusion Criteria:

* Have severe or acute back pain that limits basic movement or requires medical treatment
* History of spinal surgery or structural spine conditions (scoliosis requiring bracing/surgery)
* Have a contraindication to BFR training, identified via BFR safety screening form:
* Peripheral vascular disease (PVD)
* History of vascular surgery in arms or legs
* Skin grafts on arms or legs
* Arteriovenous fistula in limbs
* Cognitive or physical impairment that limits participation
* Hypertension or high blood pressure (uncontrolled or undiagnosed)
* Bleeding disorders (e.g., hemophilia)
* Blood clotting disorders (e.g., lupus, factor-V Leiden)
* Past history of DVT or pulmonary embolism (PE)
* Surgery in the past 12 weeks
* Recent limb immobilization (e.g., cast, boot) in the last 4 weeks
* History of stroke or transient ischemic attack (TIA)
* History of cancer
* Diagnosed heart disease
* History of rhabdomyolysis
* Diagnosed diabetes
* Sickle cell disease
* History of compartment syndrome
* History of nerve damage or injury
* Any prior complications or adverse reactions to BFR training
* Any other medical conditions that should be cleared by a physician before starting BFR
* Pregnancy(Self-reported)

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Hamstring and quadricep muscular fatigue assessment via Noraxon Electromyography | change between baseline and 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Everett Lohman, Dsc, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are not decided yet.